CLINICAL TRIAL: NCT00915785
Title: Pilot Study of 5 Azacytidine in the Treatment of Myelodysplastic Syndromes/Acute Myeloid Leukaemia With High-risk (Chromosome 7 and or Complex) Cytogenetic Abnormalities
Brief Title: Azacytidine for the Treatment of Myelodysplastic Syndromes/Acute Myeloid Leukemia (MDS/AML) With High Risk (Chromosome 7 and or Complex) Cytogenetic Abnormalities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Professor Ghulam Mufti, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05CC12; REC - 05/Q0703/168; EudraCT - 2005-003732-22
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5 azacytidine (Experimental)
  Interventions: Drug: 5 azacytidine

INTERVENTIONS:
Drug: 5 azacytidine — Patients will receive azacytidine 75 mg/m2/day SC for 7 days every 28 days for up to 6 cycles, unless they are discontinued from the treatment.

SUMMARY:
The purpose of this study is to assess the hematological and cytogenetic responses with 5 azacytidine in patients over 55 years of age with MDS/AML due to chromosome 7 abnormalities and to assess the hematological and cytogenetic response rates in patients with relapsed AML and chromosome 7 abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Abnormalities to chromosome 7, including monosomy 7 either alone or as part of a complex clone.
* Be > 55 years of age; younger if first or subsequent relapse in patient less < 55 years but with a chromosome 7 abnormality alone or as part of a complex clone.
* Have an International Prognostic Scoring System (IPSS) score of INT 1.5 and a diagnosis of RAEB or RAEB-T per French-American-British (FAB) classification criteria or a diagnosis of Myelodysplastic CMMoL per modified FAB criteria meeting the following:

  * Monocytosis in peripheral blood > 1x109/L;
  * Dysplasia in one or more myeloid cell lines;
  * 10% to 29% blasts in the BM;
  * White blood cell (WBC) < 13,000 x109/L;
* Have a life expectancy of at least 3 months;
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status Grade of 0-2.
* Have serum bilirubin levels of at least 1.5 x the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to:

  * active hemolysis (as indicated by positive direct Coombs' testing);
  * decreased or absent haptoglobin level;
  * elevated indirect bilirubin and/or lactate dehydrogenase [LDH]); or
  * ineffective erythropoiesis (as indicated by bone marrow findings).
* Have serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels of at least 2 x ULN.
* Have serum creatinine levels of at least 1.5 x ULN.
* Women of childbearing potential may participate, providing they meet the following conditions:

  * must agree to use at least 2 effective contraceptive methods throughout the study and for 3 months following the date of the last dose of study medication;
  * must have a negative serum pregnancy test obtained within 24 hours prior to Day 1.
* Males with female partners of childbearing potential must agree to use at least 2 effective contraceptive methods throughout the study and should avoid fathering a child for 6 months following the date of the last dose of study medication.
* Be able to provide written informed consent.

Exclusion Criteria:

* Prior treatment with azacitidine.
* Diagnosis of malignant disease within the previous 12 months (excluding basal cell carcinoma with no complications).
* Diagnosis of metastatic disease.
* Previous diagnosis of hepatic tumors.
* Radiation therapy, chemotherapy, or cytotoxic therapy, given to treat conditions other than MDS/AML and administered within the previous 12 months prior to the first day of treatment (Day 1).
* Known or suspected hypersensitivity to azacitidine or mannitol.
* Prior or active disease that, in the opinion of the Investigator, may interfere with the procedures or evaluations to be conducted in the study.
* Serious medical illness likely to limit survival to under or equal to 12 months after screening or likely to prevent granting of informed consent (e.g., history of severe congestive heart failure, clinically unstable cardiac disease, or pulmonary disease).
* Psychiatric illness that would prevent granting of informed consent;
* Treatment with erythropoietin or myeloid growth factors (granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor [GM-CSF]) during the previous 21 days prior to Day 1.
* Treatment with androgenic hormones during the previous 14 days prior to Day 1.
* Active viral infection with known human immunodeficiency virus (HIV) or viral hepatitis type B or C.
* Treatment with other investigational drugs within the previous 30 days prior to Day 1, or ongoing adverse events from previous treatment with investigational drugs, regardless of the time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The rate of haematological and cytogenetic response in patients with MDS/AML with a chromosome 7 abnormality either alone or as part of a complex clone | Blood - Weekly for first 2 cycles and then fortnightly. Bone marrow - Day 7 of first cycle and then 16 weekly thereafter or ealier if clinically indicated.

SECONDARY OUTCOMES:
Time to relapse after complete remission (CR) or partial remission (PR), or disease progression (per IWG criteria), censored at death | Blood - Weekly for first 2 cycles and then fortnightly. Bone marrow - Day 7 of first cycle and then 16 weekly thereafter or ealier if clinically indicated.
Duration of response and duration of improvement | Blood - Weekly for first 2 cycles and then fortnightly. Bone marrow - Day 7 of first cycle and then 16 weekly thereafter or ealier if clinically indicated.
Time to AML transformation or death from any cause | Blood - Weekly for first 2 cycles and then fortnightly. Bone marrow - Day 7 of first cycle and then 16 weekly thereafter or ealier if clinically indicated.
Additional cytogenetic markers: DNA methylation status, assessment of markers of apoptosis. Change in gene expression and single nucleotide polymorphism profiles. | Baseline, Day 7 of the first treatment cycle and then 16 weekly (or ealier if clinically indicated).

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam J Mufti, MB, DM, FRCP, FRCPath, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom